CLINICAL TRIAL: NCT00214734
Title: Evaluation of Safety, Efficacy, and Immunogenicity of ADVATE in Hemophilia A- An ADVATE Post-authorization Safety Surveillance (PASS) Study
Brief Title: ADVATE Post Authorization Safety Surveillance
Status: Completed | Type: Observational
Sponsor: Baxalta now part of Shire (Industry)
Collaborators: Baxter BioScience (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: ADVATE PASS
Record Dates: First submitted 2005-09-15; First posted 2005-09-22 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Drug: rAHF-PFM

SUMMARY:
The primary objective of this post-authorization safety surveillance is to measure the incidence of adverse events that are at least possibly related to ADVATE use, in subjects receiving ADVATE in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Subject has moderate or severe hemophilia A (baseline FVIII less than or equal to 5%)
* Subject currently has no measurable FVIII inhibitor titer greater than or equal to 1 BU (Bethesda or Nijmegen method)
* Subject has been prescribed ADVATE by their treating physician
* Subject may be of any age
* Subject or parent/legally authorized representative has provided written informed consent

Exclusion Criteria:

* None

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2004-10-14 (Actual); Study Completion 2007-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (37):
- United States (37):
  - PHOENIX CHILDRENS Hospital, Phoenix, Arizona
  - Arkansas Childrens Hospital, Little Rock, Arkansas
  - City of Hope National Medical Center, Duarte, California
  - LONG BEACH MEMORIAL MED Center, Long Beach, California
  - Children´s Hospital Los Angeles, Hemophilia Comprehensive Care Center, Division of Pediatric Hematology/Oncology, Los Angeles, California
  - Valley Children'S Hospital, Madera, California
  - Children'S Hospital of S.W. Florida, Fort Myers, Florida
  - BIODORON, Hollywood, Florida
  - Nemours Children'S Clinic, Jacksonville, Florida
  - NEMOURS CHILDREN'S CLINIC- Orlando, Orlando, Florida
  - Tampa Children'S Hospital At St. Joes, Tampa, Florida
  - University of Southern Florida, Tampa, Florida
  - Rush Presbyterian - St. Lukes Medical Center, Chicago, Illinois
  - Children´s Memorial Hospital, Chicago, Illinois
  - Indiana Hemophilia & Thrombosis Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa Regional Hemophilia Center, Department of Pediatrics, Iowa City, Iowa
  - Tulane Univ Hosp & Clinic, New Orleans, Louisiana
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - University of Michigan Med. Ctr Htc, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - PHS DEVOS CHILDRENS Hospital, Grand Rapids, Michigan
  - MUNSON MED Center, Traverse City, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - St. Louis Children'S Hospital, St Louis, Missouri
  - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Ted R. Montoya Hemophilia Treatment Center, Albuquerque, New Mexico
  - North Carolina Baptist Hospital, Hematology/Oncology Medical Center Boulevard, Winston-Salem, North Carolina
  - Phs Childrens Hosp Med Ctr Akron, Akron, Ohio
  - Children´s Hospital Medical Center Pharmacy, Hemophilia Treatment Center, Cincinnati, Ohio
  - Youngstown HTC, Youngstown, Ohio
  - Childrens Hosp of Philadelphia, Philadelphia, Pennsylvania
  - Presbyterian Medical Center, Philadelphia, Pennsylvania
  - St. Christopher´s Hospital for Children, Section of Hematology/Oncology, Philadelphia, Pennsylvania
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - Phs-So Tx Hemo Ctr-San Antonio, San Antonio, Texas
  - Children'S Hospital of the King'S Daughters, Norfolk, Virginia

REFERENCES:
- See also: To obtain more information on the study, click here/on this link. — https://clinicaltrials.takeda.com/study-detail/5f6b5fc94db2bf003ab46231